CLINICAL TRIAL: NCT05467267
Title: Personalized Urine Biomarker for Patients With Bladder Cancer: Pilot Study
Brief Title: Personalized Urine Biomarker for Patients With Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0121-21-ZIV
Record Dates: First submitted 2022-02-21; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Bladder Neoplasm
Keywords: bladder neoplasm, urine, biomarker
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor DNA - extracted from Tumor tissue and the urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TURBT — Patients with known bladder tumor undergoing TURBT - A biopsy from the tumor tissue will be taken. Peri operation a urine sample will be taken.

SUMMARY:
Introduction

Bladder cancer is the most common malignancy involving the urinary system and the ninth most common malignancy worldwide. Urothelial carcinoma is accounts for approximately 90 percent of bladder cancers in the western world.

In the United States, approximately 80,000 new cases and 17,000 deaths occur each year due to bladder cancer.

Approximately 75% of patients present with superficial disease (Ta and T1), while 25% present with muscle invasive (T2 or greater) disease. Overall, 70% of treated tumors recur, with 30% of recurrent tumors progressing to muscle invasive disease.

The majority of these patients have a recurrence after endoscopic resection, thus lifelong surveillance with periodically cystoscopy is recommended. Cystoscopy, which is the "gold standard" for the detection of bladder cancer, is an expensive and invasive procedure, and it also can miss a flat lesion, especially carcinoma in situ which is considered a high grade malignant condition, therefore better follow-up tools should be developed in order to address those issues.

Voided urinary cytology is a useful noninvasive adjunct to cystoscopy due to its high specificity, more than 90%. Although it has a high sensitivity at detecting high-grade lesions, between 80 to 90%,, in low-grade its sensitivity is very low, between 20 to 50%. Amongst the non-muscle-invasive, low grade tumors will progress to muscle-invasive or metastatic cancer at approximately 10% and roughly a third of high-grade tumors progress, therefore, close monitoring and early detection of all lesions are important for management, and noninvasive tumor markers with high accuracy for the detection of all grades of urothelial carcinoma will significantly reduce patient cost, anxiety and morbidity.

Cystoscopy in combination with cytology remains the most effective means of detecting bladder cancer. However, cystoscopy is an invasive procedure, and while cytology remains a useful method for detecting high grade tumors, its utility in detecting low grade tumors remains limited due to the lack of distinguishing cytological features between low grade disease and reactive processes. Currently there are several markers available or under investigation for the detection and monitoring/surveillance of bladder cancer, most of them have higher sensitivities, especially when used to identify low grade disease, but with lower specificities when compared to cytology. Furthermore, all of these tests must still be utilized in conjunction with cystoscopy findings.

Recently, cell-free DNA (cfDNA) isolated from urine supernatant has been shown to have great potential in bladder cancer detection and surveillance. Bladder cancer exhibits unique genetic features that can be identified from sequencing and expression of cfDNA.

Aim of study:

The aim of this study is to establish a method for a personalized urinary biomarker with the usage of well explored urothelail cancer genetic mutations in urine cfDNA, for the detection of bladder cancer presence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years old
* Able to give a written consent
* Able to provide a minimum of 60 mL of urine prior to undergoing transurethral resection of bladder tumor (TURBT)
* Presence of a bladder tumor

Exclusion Criteria:

* Active urinary infection
* Macro-hematuria
* Inadequate material for testing
* Benign bladder tumor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Study Population: The study will include 20 participants of patients with urothelial cancer of bladder who are planned for TURBT procedure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Presence of somatic mutations in bladder tumor cells | 24 months
  A set of selected somatic mutations will be checked against extracted urine cell free DNA from patients with bladder cancer, then a profile for each patient will be performed separately

IPD SHARING:
Plan to Share IPD: No